CLINICAL TRIAL: NCT04807634
Title: Role of Intravenous Lipid Emulsion in Improving Coma of Acute Antipsychotics Poisoning: A Randomized Controlled Trial in PoisonControl Center of Ain Shams University Hospitals
Brief Title: Role of Intravenous Lipid Emulsion in Improving Coma of Acute Antipsychotics Poisoning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AinShamsU RCT
Record Dates: First submitted 2021-02-10; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Coma
Keywords: Coma /antipsychotics/ lipid emulsion/acute toxicity
MeSH Terms: conditions — Coma | interventions — Fat Emulsions, Intravenous

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (RCT).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (control) (Other): Group A (control): that will receive the traditional supportive treatment for acute antipsychotic drugs overdose
  Interventions: Drug: Intravenous Lipid Emulsion (Intralipid 20%)
- Group B (case) (Other): that will receive the traditional supportive treatment for acute antipsychotic drugs overdose plus administration of 1.5 ml/kg ILE (20%) as a bolus over 1-2 minutes, followed by a continuous rate infusion of 0.25 ml/kg/min for the next 30 to 60 minutes
  Interventions: Drug: Intravenous Lipid Emulsion (Intralipid 20%)

INTERVENTIONS:
Drug: Intravenous Lipid Emulsion (Intralipid 20%) — Lipid emulsion or fat emulsion refers to an emulsion of lipid for human intravenous use. It is often referred to by the brand name of the most commonly used version, Intralipid, which is an emulsion of soy bean oil, egg phospholipids and glycerin, and is available in 10%, 20% and 30% concentrations. The 30% concentration is not approved for direct intravenous infusion, but should be mixed with amino acids and dextrose as part of a total nutrient admixture.
  Other Names: Intralipid 20%

SUMMARY:
Intravenous Lipid Emulsion in Improving Coma Of Antipsychotic drugs Acute Poisoning: A Randomized Controlled Trial in Poison Control Center of Ain Shams University Hospitals

DETAILED DESCRIPTION:
Intravenous lipid emulsions (ILEs) have been recently used in treatment of acute toxicity caused by lipophilic drugs including local anesthetics, antidepressants, anti-arrhythmics, beta blockers and calcium channel antagonists with few case reports concerning their use in treatment of acute antipsychotics overdose (Muller et al., 2015).

To the best of our knowledge, no randomized controlled trials (RCTs) have been performed to evaluate the antidotal effect of ILEs on the level of consciousness of acutely poisoned patients by antipsychotics and their routine metabolic profile tests.

Acute poisoning by antipsychotics could result in various life-threatening toxic effects mainly on cardiovascular and central nervous systems (CNS). Tachycardia, hypotension, and QT prolongation in electrocardiogram are the most common cardiovascular findings while sedation, extrapyramidal symptoms, agitation, and coma are the most common CNS findings following acute antipsychotic exposures (Divac et al., 2014).

As acute antipsychotic drugs overdose lack specific antidote, the primary goal in treatment is aggressive supportive therapy. In order to prevent CNS depression and respiratory failure, patients may need to be supported by mechanical ventilation. Hypotension is treated by intravenous fluids with use of direct-acting vasopressors (Orazel et al., 2019).

Several mechanisms for the antidotal properties of ILEs have been proposed including their ability to capture lipophilic drugs and extract them from vital organs such as the heart and brain thus reducing their toxicity, preferential distribution of lipophilic drugs into a circulating lipid phase, thereby reducing tissue drug concentrations. In addition, ILEs have direct inotropic effect due to improved fatty acid oxidative metabolism resulting in restoration of myocardial contractility (Zyoud et al., 2016 & Kehayova et al., 2019).

Sample size:

• Based on the calculated sample size by statistics committee (Community Medicine, Environmental, and Occupational Medicine Department - Faculty of Medicine, Ain shams University), a total of at least 30 patients with history of acute intoxication by antipsychotic drugs will be enrolled and randomly assigned into case (n=15) and control (n=15) groups.

Method of rondamization:

• Randomization will be achieved via a computer-generated random -sequence table.

On admission, the patient will receive the conventional management including history taking, clinical examination, investigations and treatment .

Examination will be repeated every six hours through the period of hospital stay of the patient.

All clinical data of the patient will be recorded in a special sheet that include the following data :

1. Sociodemographic data:

   * Age.
   * Gender.
   * Residence
2. Intoxication data:

   * Type of antipsychotic drug responsible for intoxication.
   * Amount of antipsychotic drug (if available).
   * Mode of poisoning, whether suicidal, accidental, criminal or therapeutic error.
   * Route of intake of the poison.
   * Time elapsed between the exposure and arrival to the PCC-ASU (delay time).
   * Preconsultation management.
   * Presence of comorbidities (as underlying medical or psychiatric diseases).
   * The current medications used by the patient including all drugs used in treatment of diseases.
3. Clinical data (on admission and during hospital stay):

   * In both groups, detailed examination of the patients will be carried out on admission and routinely according to the severity of poisoning.
   * Assessment of the level of consciousness of all patients under the study will be carried out on admission and every six hours by using Glasgow coma scale (GCS) and Alert, Voice, Pain, Unresponsive (AVPU) scale till the patient discharge or mortality.
4. Investigations:

   * Laboratory: all required laboratory investigations will be performed including arterial blood gas (ABG) analysis, and routine metabolic profile tests (e.g. glucose, sodium, potassium, urea and creatinine).
   * Other required investigations: Electrocardigraphy (ECG) will be done on admission and 12 h later, then every 24 h till the patient discharge or mortality.

ELIGIBILITY:
Inclusion Criteria:

* All adult comatose patients admitted to the ICU of Poison Control Center of Ain Shams University Hospitals with positive history of antisychotic drugs overdose during the period starting from the beginning of March 2020 to the end of Septemper 2021

Exclusion Criteria:

* Based on the possibility of heterogeneity in hemodynamic parameters, laboratory variables, GCS and/or AVPU Scale, the following patients will be excluded:

  * Patients less than 18 years and more than 65 years.
  * Pregnant and lactating females.
  * Co-ingestion of other agents.
  * Presence of medical diseases (e.g. renal, hepatic, cardiovascular diseases) and chronic pancreatitis.
  * History of head trauma.
  * Presence of conditions where ILE is contraindicated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Complete recovery | 6 months
  Regaining consciousness with galasco coma scale 15/15 without presence of other clinical manifestations denoting antipsychotics toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Manal A Abdel Salam, Professor, Study Chair — Ain Shams University
Locations (1):
- Hend salama shalby El Far, Cairo, Egypt

REFERENCES:
- [Background] Berling I, Buckley NA, Isbister GK. The antipsychotic story: changes in prescriptions and overdose without better safety. Br J Clin Pharmacol. 2016 Jul;82(1):249-54. doi: 10.1111/bcp.12927. Epub 2016 Apr 15. PMID 26945707
- [Background] Divac N, Prostran M, Jakovcevski I, Cerovac N. Second-generation antipsychotics and extrapyramidal adverse effects. Biomed Res Int. 2014;2014:656370. doi: 10.1155/2014/656370. Epub 2014 Jun 3. PMID 24995318
- [Background] Levine M, Ruha AM. Overdose of atypical antipsychotics: clinical presentation, mechanisms of toxicity and management. CNS Drugs. 2012 Jul 1;26(7):601-11. doi: 10.2165/11631640-000000000-00000. PMID 22668123
- [Background] Muller SH, Diaz JH, Kaye AD. Clinical applications of intravenous lipid emulsion therapy. J Anesth. 2015 Dec;29(6):920-6. doi: 10.1007/s00540-015-2036-6. Epub 2015 Jun 7. PMID 26049929
- [Background] Zyoud SH, Waring WS, Al-Jabi SW, Sweileh WM, Rahhal B, Awang R. Intravenous Lipid Emulsion as an Antidote for the Treatment of Acute Poisoning: A Bibliometric Analysis of Human and Animal Studies. Basic Clin Pharmacol Toxicol. 2016 Nov;119(5):512-519. doi: 10.1111/bcpt.12609. Epub 2016 May 20. PMID 27098056